CLINICAL TRIAL: NCT07086989
Title: Cardiovascular Risk in Children With Chronic Conditions Study
Acronym: CR3C
Status: Recruiting | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Kiss Tamás, Principal Investigator, Semmelweis University
Other Study IDs: NNGYK/00994-4/2025
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Kidney Transplant; Familial Hypercholesterolaemia; Type 1 Diabetes Mellitus (T1DM); Type 2 Diabetes Mellitus (T2DM); Chronic Kidney Disease; Kawasaki Disease; Liver Transplant; Obesity and Overweight; Hypertension; Coarctation of Aorta; Bone Marrow Transplant; Cancer (Solid Tumors); Leukemia; Lymphoma; Lipoprotein(a); Aorta Stenosis; Non Alcoholic Fatty Liver Disease; Dyslipaemia; White Coat Hypertension; Pulmonary Hypertension; Juvenile Idiopahtic Arthritis; Systemic Lupus Erthematosus; Inflammatory Bowel Disease (IBD); HIV Infection; Transposition of Great Arteries
Keywords: cardiovascular risk; vasculature; children with chronic conditions
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Mucocutaneous Lymph Node Syndrome; Obesity; Overweight; Hypertension; Aortic Coarctation; Neoplasms; Leukemia; Lymphoma; Aortic Valve Stenosis; Non-alcoholic Fatty Liver Disease; White Coat Hypertension; Hypertension, Pulmonary; Inflammatory Bowel Diseases; HIV Infections; Transposition of Great Vessels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum and blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children living with chronic health conditions face a higher risk of developing cardiovascular diseases than their peers, largely due to the accelerated aging of the heart and blood vessels. Although experts recognize this elevated risk and recommend close monitoring and early intervention, the underlying mechanisms driving this phenomenon remain poorly understood. At present, no effective interventions specifically target its root causes.

Recent research shows that both large blood vessels (such as the carotid artery) and small vessels (such as those in the retina) can display early signs of damage decades before clinically apparent heart or vascular disease emerges. This accelerated vascular aging can result from multiple factors - including disease-related processes such as persistent inflammation and metabolic disturbances, treatment-related effects such as chemotherapy or long-term steroid use, and lifestyle changes associated with chronic illness, such as reduced physical activity and altered eating habits. However, it is still unclear how these factors influence the development and progression of vascular changes in children as they grow. Importantly, these changes can be monitored through non-invasive methods, offering a unique opportunity to study at-risk patients many years before overt cardiovascular disease develops.

Identifying these early changes may enable us to detect and track individuals at heightened risk well in advance of clinical disease. This study aims to deepen our understanding of the causes of increased cardiovascular risk in children with chronic conditions and to lay the groundwork for earlier, more targeted prevention strategies.

ELIGIBILITY:
Inclusion criteria:

1. Individuals aged between 6 and 25 years;
2. Diagnosed with a chronic childhood condition/disease associated with an increased risk of early cardiovascular disease;
3. Provided informed consent (if over 18 years old) or had informed consent provided by their legal guardian (if under 18 years old) following appropriate information about the study.

Chronic childhood conditions/diseases associated with increased risk of early cardiovascular disease are defined according to the 2019 American Heart Association recommendations (https://doi.org/10.1161/CIR.0000000000000618), as well as other conditions/diseases for which at least two large-scale epidemiological studies have demonstrated an increased risk of cardiovascular disease.

Exclusion criteria:

1. Severe intellectual and developmental disability;
2. Decompensated heart failure;
3. Severe primary immunodeficiency;
4. Ongoing intravenous chemotherapy;
5. Infectious diseases posing a public health risk; or
6. History of regular alcohol or drug use.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, adolescents, and young adults (aged 6-25 years) who have been diagnosed with a chronic childhood condition associated with an increased risk of early-onset cardiovascular disease, and who are receiving care at a university-affiliated clinical setting. Participants must be capable of providing informed consent (if ≥18 years old) or have consent provided by a legal guardian (if <18 years old). The population excludes individuals with severe intellectual disabilities, decompensated heart failure, severe primary immunodeficiencies, active intravenous chemotherapy, communicable diseases that pose a public health risk, or a history of regular alcohol or drug use.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness | At baseline and at the time of annual follow-up
  Assessed by carotid-femoral pulse wave velocity
Endothelial function of the brachial artery | At baseline and at the time of annual follow-up
  Evaluated using flow-mediated dilation measured by ultrasound
Retinal vessel diameter | At baseline and at the time of annual follow-up
  Assessed by static retinal vessel analysis
Retinal vessel fractal dimension and tortuosity | At baseline and at the time of annual follow-up
  Assessed by static retinal vessel analysis

SECONDARY OUTCOMES:
Endothelial function in capillaries | At baseline and at the time of annual follow-up
  Assessed by flow-mediated dilation using laser speckle contrast imaging
Retinal neurovascular coupling | At baseline and at the time of annual follow-up
  Assessed by dynamic retinal vessel analysis

CONTACTS AND LOCATIONS:
Overall Officials: Tamas Kiss, MD, PhD, Principal Investigator — Semmelweis University, Pediatric Center
Locations (3):
- Hungary (3):
  - Semmelweis University, Department of Surgery, Transplantation and Gastroenterology, Budapest
  - Semmelweis University, Pediatric Center, Budapest
  - Semmelweis University, Institute of Preventive Medicine and Public Health, Budapest

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hanssen H, Moholdt T, Bahls M, Biffi A, Siegrist M, Lewandowski AJ, Biondi-Zoccai G, Cavarretta E, Kokkvoll A, Lochen ML, Maestrini V, Pinto RS, Palermi S, Thivel D, Wojcik M, Hansen D, Van Craenenbroeck EM, Weghuber D, Kraenkel N, Tiberi M. Lifestyle interventions to change trajectories of obesity-related cardiovascular risk from childhood onset to manifestation in adulthood: a joint scientific statement of the task force for childhood health of the European Association of Preventive Cardiology and the European Childhood Obesity Group. Eur J Prev Cardiol. 2023 Oct 10;30(14):1462-1472. doi: 10.1093/eurjpc/zwad152. PMID 37491406
- [Background] Varley BJ, Nasir RF, Skilton MR, Craig ME, Gow ML. Early Life Determinants of Vascular Structure in Fetuses, Infants, Children, and Adolescents: A Systematic Review and Meta-Analysis. J Pediatr. 2023 Jan;252:101-110.e9. doi: 10.1016/j.jpeds.2022.08.033. Epub 2022 Aug 24. PMID 36029824
- [Background] Raitakari O, Pahkala K, Magnussen CG. Prevention of atherosclerosis from childhood. Nat Rev Cardiol. 2022 Aug;19(8):543-554. doi: 10.1038/s41569-021-00647-9. Epub 2022 Jan 5. PMID 34987194
- [Background] de Ferranti SD, Steinberger J, Ameduri R, Baker A, Gooding H, Kelly AS, Mietus-Snyder M, Mitsnefes MM, Peterson AL, St-Pierre J, Urbina EM, Zachariah JP, Zaidi AN. Cardiovascular Risk Reduction in High-Risk Pediatric Patients: A Scientific Statement From the American Heart Association. Circulation. 2019 Mar 26;139(13):e603-e634. doi: 10.1161/CIR.0000000000000618. PMID 30798614
- [Background] Jacobs DR Jr, Woo JG, Sinaiko AR, Daniels SR, Ikonen J, Juonala M, Kartiosuo N, Lehtimaki T, Magnussen CG, Viikari JSA, Zhang N, Bazzano LA, Burns TL, Prineas RJ, Steinberger J, Urbina EM, Venn AJ, Raitakari OT, Dwyer T. Childhood Cardiovascular Risk Factors and Adult Cardiovascular Events. N Engl J Med. 2022 May 19;386(20):1877-1888. doi: 10.1056/NEJMoa2109191. Epub 2022 Apr 4. PMID 35373933
- [Background] Townsend N, Kazakiewicz D, Lucy Wright F, Timmis A, Huculeci R, Torbica A, Gale CP, Achenbach S, Weidinger F, Vardas P. Epidemiology of cardiovascular disease in Europe. Nat Rev Cardiol. 2022 Feb;19(2):133-143. doi: 10.1038/s41569-021-00607-3. Epub 2021 Sep 8. PMID 34497402